CLINICAL TRIAL: NCT01718691
Title: Phase II Clinical Study of SyB L-0501 in Combination With Rituximab in Patients With Untreated, Low-grade B-cell Non-Hodgkin's Lymphoma and Mantle Cell Lymphoma (Multicenter, Open-label).
Brief Title: Efficacy and Safety Study of SyB L-0501 in Combination With Rituximab in Patients With Untreated, Low-grade B Cell Non-Hodgkin's Lymphoma and Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011002
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Results first posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-03

CONDITIONS: Low-grade B Cell Non-Hodgkin's Lymphoma; Mantle Cell Lymphoma Where Hematopoietic Stem Cell Transplantation is Not Indicated
MeSH Terms: interventions — Rituximab

ARMS (1):
- SyB L-0501＋rituximab (Experimental)
  Interventions: Drug: SyB L-0501; Drug: rituximab

INTERVENTIONS:
Drug: SyB L-0501 — A dose of 90 mg/m^2/day of SyB L-0501 is administered on Day 1 and Day 2 as an IV drip infusion, followed by 26-day observation. This is 1 cycle (28 days), which will be repeated for a maximum of 6 times.
Drug: rituximab — A dose of 375 mg/m^2 of rituximab is administered on Day 1 (Day 0 in Cycle 1 only) as an IV drip infusion, followed by 26-day observation. This is 1 cycle (28 days), which will be repeated for a maximum of 6 times. From Cycle 2, rituximab will be coadministered with SyB L-0501 on Day 1. However, if the investigator or sub-investigator judges that the coadministration is difficult, rituximab may be administered on Day 0.

SUMMARY:
The purpose of this study is to assess the efficacy and safety of SyB L-0501 (two-day consecutive 90 mg/m2/day IV drip infusions) in combination with rituximab (375 mg/m2 IV drip infusion) on untreated, low-grade B cell non-Hodgkin's lymphoma and mantle cell lymphoma where hematopoietic stem cell transplantation is not indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are histopathologically confirmed to have the following cluster of differentiation 20 (CD20) positive low-grade B cell non-Hodgkin's lymphoma or mantle cell lymphoma by lymph node biopsy or evaluable tissue biopsy within 6 months before the registration WHO Classification of Tumors (fourth edition):

   * Small lymphocytic lymphoma
   * Splenic marginal zone B-cell lymphoma
   * Lymphoplasmacytic lymphoma
   * Extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue (MALT lymphoma)
   * Nodal marginal zone B-cell lymphoma
   * Follicular lymphoma (Grade 1, 2, 3a)
   * Mantle cell lymphoma
2. Patients with a measurable lesion ( > 1.5 cm in major axis on CT)
3. Patients without a medical history
4. Patients with at least 1 of the following clinical symptoms or signs (excluding mantle cell lymphoma):

   * Bulky disease measuring > 7 cm in major axis on CT (excluding spleen)
   * B symptoms

     1. Fever exceeding 38.0ºC of unknown cause
     2. Night sweats
     3. Weight decrease exceeding 10% within 6 months before patient registration
   * Elevated serum LDH or beta 2 microglobulin
   * Three or more regional lymph nodes of > 3 cm in major axis on CT
   * Symptomatic splenomegaly
   * Intracranial pressure
   * Pleural effusion/ascites retention
5. Patients expected to live for at least 3 months
6. Patients aged between 20 and 79 years (at the time of registration)
7. Patients whose Eastern Cooperative Oncology Group (ECOG) performance status (P.S.) is 0～2
8. Patients with adequately maintained major organ function (bone marrow, heart, lungs, liver, kidneys)

   * Neutrophil count: not less than 1,500 /mm3
   * Platelet count: not less than 75,000 /mm3
   * Aspartate aminotransferase (AST)[Glutamic oxaloacetic transaminase (GOT)]: not more than 3 times the standard upper limit for the site
   * Alanine aminotransferase (ALT)[Glutamic pyruvic transaminase (GPT)]: not more than 3 times the standard upper limit for the site
   * Total bilirubin: not more than 1.5 times the standard upper limit for the site
   * Serum creatinine: not more than 1.5 times the standard upper limit for the site
   * Arterial partial pressure of oxygen (PaO2): not less than 65 mmHg
   * Electrocardiogram shows no abnormal findings that require treatment
   * Echocardiogram of left ventricular ejection fraction (LVEF): not less than 55%
9. Patients whose informed consent has been obtained in person

Exclusion Criteria:

Patients who fall under any one of the following criteria are to be excluded

1. Patients whose transformation has been confirmed histopathologically
2. Mantle cell lymphoma patients aged 65 years or younger
3. Patients who were administered or received transfusion of cytokine formulations such as G-CSF (granulocyte colony stimulating factor) and erythropoietin within 14 days before pre-registration test
4. Patients with severe active infectious disorders (receiving antibiotics, antifungals, or antivirus IV injection)
5. Patients with serious complications (such as hepatic or renal failure)
6. Patients with severe complications of cardiac disease (examples: myocardial infarction, ischemic heart disease) or its previous history within 2 years before patient registration, and patients with arrhythmia requiring a treatment
7. Patients with serious gastrointestinal conditions (persistent or severe nausea/vomiting or diarrhea)
8. Patients who are positive for hepatitis B surface (HBs) antigen, hepatitis C virus (HCV) antibody or HIV antibody [if HBs or hepatitis B core (HBc) positive, patients whose hepatitis B virus (HBV)-DNA test results indicate positive]
9. Patients with serious bleeding tendencies [such as disseminated intravascular coagulation (DIC)]
10. Patients having or suspected of having symptoms indicative of the central nervous system (CNS) involvement
11. Patients with interstitial pneumonitis, pulmonary fibrosis, pulmonary emphysema complications requiring treatment or its medical history.
12. Patients with active multiple primary cancer
13. Patients who received chemotherapy, radiotherapy, antibody therapy and antitumor steroid therapy in the past
14. Patients with complications or medical history of autoimmune haemolytic anaemia
15. Patients who were administered investigative or unapproved drugs within 3 months before patient registration
16. Patients with addiction to drugs or narcotics, or alcoholism
17. Patients who have previously received hematopoietic stem cell transplantation
18. Patients who are or may be pregnant, lactating patients
19. Patients, whether male or female, who do not agree to use contraception
20. Patients otherwise judged by the investigator or the sub-investigator to be unsuitable for inclusion in the study

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- Japan (14):
  - Research site, Nagoya, Aichi-ken
  - Research site, Kashiwa, Chiba
  - Research site, Fukuoka, Fukuoka
  - Research site, Sapporo, Hokkaido
  - Research site, Kagoshima, Kagoshima-ken
  - Research site, Isehara, Kanagawa
  - Research site, Kyoto, Kyoto
  - Research site, Sendai, Miyagi
  - Research site, Nagasaki, Nagasaki
  - Research site, Moriguchi, Osaka
  - Research site, Izumo, Shimane
  - Research site, Hamamatsu, Shizuoka
  - Research site, Utsunomiya, Tochigi
  - Research site, Tokyo, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- Low-grade B-cell Non-Hodgkin's Lymphoma: Subjects in the SyB L-0501＋ rituximab arm with primary disease of Low-grade B-cell non-Hodgkin's lymphoma.
- Mantle Cell Lymphoma: Subjects in the SyB L-0501＋ rituximab arm with primary disease of Mantle cell lymphoma.
Period: Overall Study
Arm/Group | Low-grade B-cell Non-Hodgkin's Lymphoma | Mantle Cell Lymphoma
Started | 60 | 10
Completed | 42 | 9
Not Completed | 18 | 1

BASELINE CHARACTERISTICS:
Population: Of the 70 subjects enrolled, one who did not receive the investigational product was excluded. Therefore, the total number of Baseline Participants is 69.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-grade B-cell Non-Hodgkin's Lymphoma | Mantle Cell Lymphoma | Total
Number analyzed (Participants) | 59 | 10 | 69
Age, Customized [Number; unit: participants]
  ˂65 years | 36 | 0 | 36
  ≥65 years | 23 | 10 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 1 | 38
  Male | 22 | 9 | 31
Performance status (ECOG scale) [Number; unit: participants] — The criteria of Eastern Cooperative Oncology Group (ECOG) performance status are shown below.
  0: Symptoms are absent, no restrictions on lifestyle
  1. Symptoms are present; no restrictions on walking; Strenuous physical activity is restricted
  2. Symptoms are present; able to walk; able to perform self-care; Spends over 50% of waking hours out of bed
  participants
    0 | 42 | 7 | 49
    1 | 16 | 3 | 19
    2 | 1 | 0 | 1
Diagnosis (WHO classification) [Number; unit: participants]
  Small lymphocytic lymphoma | 2 | 0 | 2
  Lymphoplasmacytic lymphoma | 2 | 0 | 2
  Splenic marginal zone lymphoma | 0 | 0 | 0
  B-EMZL(MALT lymphoma) | 4 | 0 | 4
  Nodal marginal zone B-cell lymphoma | 0 | 0 | 0
  Follicular lymphoma | 51 | 0 | 51
  Mantle cell lymphoma | 0 | 10 | 10
Clinical stage (Ann Arbor staging classification) [Number; unit: participants] — The criteria of Ann Arbor staging classification are shown below.
  I: Invasion of 1 lymph node region II: Invasion of 2 or more lymphatic regions confined to 1 side of the diaphragm III: Invasion of multiple lymph node regions spanning above and below the diaphragm IV: Diffuse invasion to an organ or area other than 1 or multiple lymphatic tissues, regardless of the presence/absence of lymph node lesions.
  participants
    I - II | 15 | 0 | 15
    III | 9 | 0 | 9
    IV | 35 | 10 | 45
Number of lymph node regions [Number; unit: participants]
  0 region | 0 | 0 | 0
  1 region | 12 | 1 | 13
  2 regions | 6 | 1 | 7
  3 regions | 4 | 2 | 6
  4 regions or more | 37 | 6 | 43
Number of extranodal lesions [Number; unit: participants]
  0 - 1 lesion | 50 | 4 | 54
  2 or more lesions | 9 | 6 | 15
Tumor diameter (1) [Number; unit: participants]
  ≥5 cm | 38 | 4 | 42
  ˂5 cm | 21 | 6 | 27
Tumor diameter (2) [Number; unit: participants]
  ≥7 cm | 28 | 1 | 29
  ˂7 cm | 31 | 9 | 40
Lactate dehydrogenase (LDH) [Number; unit: participants]
  ≤ upper limit of normal range | 45 | 7 | 52
  High | 14 | 3 | 17
Beta 2 microglobulin [Number; unit: participants]
  ≤ upper limit of normal range | 15 | 3 | 18
  High | 44 | 7 | 51
C-reactive protein (CRP) [Number; unit: participants]
  ≤ upper limit of normal range | 39 | 8 | 47
  High | 20 | 2 | 22
Hepatomegaly [Number; unit: participants]
  Yes | 3 | 1 | 4
  No | 56 | 9 | 65
Splenomegaly [Number; unit: participants]
  Yes | 19 | 0 | 19
  No | 40 | 10 | 50
Enlarged kidney [Number; unit: participants]
  Yes | 1 | 0 | 1
  No | 58 | 10 | 68
B symptoms (fever) [Number; unit: participants]
  Yes | 0 | 0 | 0
  No | 59 | 10 | 69
B symptoms (night sweats) [Number; unit: participants]
  Yes | 3 | 0 | 3
  No | 56 | 10 | 66
B symptoms (weight loss) [Number; unit: participants]
  Yes | 2 | 0 | 2
  No | 57 | 10 | 67
Symptomatic splenomegaly [Number; unit: participants]
  Yes | 5 | 0 | 5
  No | 54 | 10 | 64
Pressure symptoms [Number; unit: participants]
  Yes | 14 | 0 | 14
  No | 45 | 10 | 55
Pleural effusion/ascites retention [Number; unit: participants]
  Yes | 5 | 0 | 5
  No | 54 | 10 | 64
Bone marrow invasion [Number; unit: participants]
  Positive | 34 | 8 | 42
  Negative | 24 | 2 | 26
  Undetermined | 1 | 0 | 1
Chromosome abnormality [Number; unit: participants]
  Yes | 13 | 4 | 17
  No | 43 | 5 | 48
  Unknown | 3 | 1 | 4
Previous medical history [Number; unit: participants]
  Yes | 31 | 7 | 38
  No | 28 | 3 | 31
Concomitant disease [Number; unit: participants]
  Yes | 53 | 10 | 63
  No | 6 | 0 | 6
FLIPI risk category [Number; unit: participants] — The criteria for Follicular Lymphoma International Prognostic Index (FLIPI) are shown below.
  * Low: No or 1 poor prognostic factor(s)
  * Intermediate: 2 poor prognostic factors
  * High: 3-5 poor prognostic factors
  participants
    Low | 17 | NA — The subjects with mantle cell lymphoma were not included in this examination. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Intermediate | 24 | NA — The subjects with mantle cell lymphoma were not included in this examination. | NA — Total not calculated because data are not available (NA) in one or more arms.
    High | 18 | NA — The subjects with mantle cell lymphoma were not included in this examination. | NA — Total not calculated because data are not available (NA) in one or more arms.
IPI risk category [Number; unit: participants] — The criteria for International Prognostic Index are shown below.
  * Low: 0 or 1poor prognostic factors
  * Intermediate (Low): 2 poor prognostic factors
  * Intermediate (High): 3 poor prognostic factors
  * High: 4 or 5 poor prognostic factors
  participants
    Low | 27 | 0 | 27
    Intermediate (Low) | 21 | 2 | 23
    Intermediate (High) | 10 | 7 | 17
    High | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate (CR + CRu) Based on International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphomas (1999)(IWRC)
Description: The criteria for CR and CRu based on IWRC are shown below.
  CR: Fulfills all of the following
  * Disappearance of all detectable disease
  * LN* > 1.5 cm must decrease to ≤ 1.5 cm
  CRu: Fulfills all of the following
  * LN >1.5 cm; SPD** decrease >75%
  * indeterminate bone marrow
    * LN: lymph nodes or nodal masses ** SPD: sum of the products of the greatest diameters
Time Frame: Up to 30 weeks
Measure: Number; unit: percentage of participants
Groups:
- Total: All subjects in the SyB L-0501＋ rituximab arm
Arm/Group | Low-grade B-cell Non-Hodgkin's Lymphoma | Mantle Cell Lymphoma | Total
Number analyzed (Participants) | 59 | 10 | 69
percentage of participants | 67.8 | 70.0 | 68.1

2. Secondary Outcome: Overall Response Rate (Antitumor Effect: PR or Better) Based on International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphomas (1999)(IWRC)
Description: The criteria for PR based on IWRC are shown below.
  PR: SPD regressed > 50%
Time Frame: Up to 30 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Low-grade B-cell Non-Hodgkin's Lymphoma | Mantle Cell Lymphoma | Total
Number analyzed (Participants) | 59 | 10 | 69
percentage of participants | 96.6 | 90.0 | 95.7

3. Secondary Outcome: Complete Response Rate (CR) Based on Revised Response Criteria for Malignant Lymphoma (2007)(Revised RC)
Description: The criteria for CR based on the Revised RC are shown below.
  Definition: Disappearance of all evidence of disease
  Nodal Masses:
  1. [18F]fluorodeoxyglucose (FDG)-avid or PET positive prior to therapy; mass of any size permitted if PET negative.
  2. Variably FDG-avid or PET negative; regression to normal size on CT.
  Spleen, Liver:
  Not palpable, nodules disappeared
  Bone Marrow:
  Infiltrate cleared on repeat biopsy; if indeterminate by morphology, immunohistochemistry should be negative.
Time Frame: Up to 30 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Low-grade B-cell Non-Hodgkin's Lymphoma | Mantle Cell Lymphoma | Total
Number analyzed (Participants) | 59 | 10 | 69
percentage of participants | 64.4 | 80.0 | 66.7

4. Secondary Outcome: Overall Response Rate (PR or Better) Based on Revised Response Criteria for Malignant Lymphoma (2007)(Revised RC)
Description: The criteria for PR based on the Revised RC are shown below.
  Definition: Regression of measurable disease and no new sites
  Nodal Masses:
  50% or more decrease in SPD of up to 6 largest dominant masses; no increase in size of other nodes
  1. FDG-avid or PET positive prior to therapy; one or more PET positive at previously involved site
  2. Variably FDG-avid or PET negative; regression on CT
  Spleen, Liver:
  50% or more decrease in SPD of nodules (for single nodule in greatest transverse diameter); no increase in size of liver or spleen
  Bone Marrow:
  Irrelevant if positive prior to therapy; cell type should be specified.
Time Frame: Up to 30 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Low-grade B-cell Non-Hodgkin's Lymphoma | Mantle Cell Lymphoma | Total
Number analyzed (Participants) | 59 | 10 | 69
percentage of participants | 96.6 | 90.0 | 95.7

5. Secondary Outcome: Complete Response Rate Based on WHO Handbook for Reporting Results of Cancer Treatment (1979)
Description: The criteria for Complete response based on WHO Handbook for Reporting Results of Cancer Treatment (1979) are shown below.
  Measurable disease:
  The disappearance of all known disease, determined by 2 observations not less than 4 weeks apart.
  Unmeasurable disease:
  Complete disappearance of all known disease for at least 4 weeks.
  Bone metastases:
  Complete disappearance of all lesions on X-ray or scan for at least 4 weeks.
Time Frame: Up to 30 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Low-grade B-cell Non-Hodgkin's Lymphoma | Mantle Cell Lymphoma | Total
Number analyzed (Participants) | 59 | 10 | 69
percentage of participants | 22.0 | 40.0 | 24.6

6. Secondary Outcome: Overall Response Rate (PR or Better) Based on "WHO Handbook for Reporting Results of Cancer Treatment (1979)"
Description: The criteria for Overall response rate (PR or better) based on "WHO Handbook for Reporting Results of Cancer Treatment (1979)" are shown below.
  Definition of PR:
  Measurable disease:
  50% or more decrease in total tumor size of the lesions which have been measured to determine the effect of therapy by 2 observations not less than 4 weeks apart. In addition there can be no appearance of new lesions or progression of any lesion.
  Unmeasurable disease:
  Estimated decrease in tumor size of 50% or more for at least 4 weeks.
  Bone metastases:
  Partial decrease in size of lytic lesions, recalcification of lytic lesions, or decreased density of blastic lesions for at least 4 weeks.
Time Frame: Up to 30 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Low-grade B-cell Non-Hodgkin's Lymphoma | Mantle Cell Lymphoma | Total
Number analyzed (Participants) | 59 | 10 | 69
percentage of participants | 86.4 | 90.0 | 87.0

7. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is the period from registration date to the earliest onset date of any progression event calculated using the Kaplan-Meier estimator. The median and the 95% confidence interval (CI) were calculated using Greenwood's formula.
  Progression event was defined as progression (includes recurrence/relapse), initiation of post-study treatment, confirmation of other malignant tumor, or death due to any given cause. The date of progression was determined based on overall response assessed using IWRC, Revised RC, and WHO, and assessment by the primary physicians (excluding overall response).
Time Frame: Up to 30 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Low-grade B-cell Non-Hodgkin's Lymphoma | Mantle Cell Lymphoma | Total
Number analyzed (Participants) | 59 | 10 | 69
days | NA [654.0 to NA] — The PFS rate during this observation period was 57.7%, which was higher than 50% and therefore, 50% PFS could not be calculated. | NA [NA to NA] — The PFS rate during this observation period was 57.7%, which was higher than 50% and therefore, 50% PFS could not be calculated. | NA [654.0 to NA] — The PFS rate during this observation period was 57.7%, which was higher than 50% and therefore, 50% PFS could not be calculated.

8. Secondary Outcome: Duration of Response (DOR)
Description: DOR is the period from the date of achieving CR, CRu or PR in the responders to the earliest onset date of any progression events calculated using the Kaplan-Meier estimator. The median and the 95% CI were calculated using Greenwood's formula.
  The date of achieving CR, CRu or PR was determined based on the overall response assessed using IWRC. The date of progression was determined based on overall response assessed using IWRC, Revised RC and WHO, and assessment by the primary physicians (excluding overall response).
  Progression event was defined as progression (includes recurrence/relapse), initiation of post-study treatment, confirmation of other malignant tumor, or death due to any given cause.
Time Frame: Up to 30 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Low-grade B-cell Non-Hodgkin's Lymphoma | Mantle Cell Lymphoma | Total
Number analyzed (Participants) | 59 | 10 | 69
days | NA [541.0 to NA] — Because response was maintained in most subjects (of 66 subjects assessed as PR or better in the overall response assessment, eleven experienced a progression event). | NA [NA to NA] — Because response was maintained in most subjects (of 66 subjects assessed as PR or better in the overall response assessment, eleven experienced a progression event). | NA [541.0 to NA] — Because response was maintained in most subjects (of 66 subjects assessed as PR or better in the overall response assessment, eleven experienced a progression event).

9. Secondary Outcome: Overall Survival (OS)
Description: Death due to any given cause was defined as an event. OS was calculated using the Kaplan-Meier estimator. The median and the 95% CI were calculated using Greenwood's formula.
Time Frame: Up to 30 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Low-grade B-cell Non-Hodgkin's Lymphoma | Mantle Cell Lymphoma | Total
Number analyzed (Participants) | 59 | 10 | 69
days | NA [NA to NA] — Because no event of death occurred. | NA [NA to NA] — Because no event of death occurred. | NA [NA to NA] — Because no event of death occurred.

10. Secondary Outcome: Number of Subjects With Adverse Event, Related Adverse Event, Serious Adverse Event, and Discontinuation Due to Adverse Event
Description: Adverse events were evaluated using Common Terminology Criteria for Adverse Events (CTCAE) v4.0, Japan Clinical Oncology Group/Japan Society of Clinical Oncology (JCOG/JSCO) version, and were encoded using Medical Dictionary for Regulatory Activities (MedDRA) Ver.16.1.
Time Frame: up to 30 weeks
Measure: Number; unit: participants
Arm/Group | Total
Number analyzed (Participants) | 69
participants
  Any adverse event | 69
  Adverse drug reaction | 69
  SAE | 9
  Death | 0
  Discontinuation due to adverse events | 0

11. Secondary Outcome: Laboratory Test Abnormalities (Biochemical Tests)
Description: Abnormalities in laboratory test values in overall study period were analyzed. Severity of abnormalities were evaluated using CTCAE. Grade 1 : mild Grade 2 : moderate Grade 3 : severe or medically significant but not immediately life-threatening Grade 4 : life threatening or disabling Grade 5 : death related to AE
Time Frame: up to 30 weeks
Measure: Number; unit: participants
Arm/Group | Total
Number analyzed (Participants) | 69
participants
  Grade 3 : AST(GOT) | 3
  Grade 3 : ALT(GPT) | 3
  Grade 3 : γ-GTP | 1
  Grade 4 : Uric acid | 1
  Grade 3 : Na decrease | 1
  Grade 3 : K decrease | 2
  Grade 3 : K increase | 1

12. Secondary Outcome: Laboratory Test Abnormalities (Hematology Tests)
Description: as for outcome 11
Time Frame: up to 30 weeks
Measure: Number; unit: participants
Arm/Group | Total
Number analyzed (Participants) | 69
participants
  Grade 3 : White blood cell count decreased | 45
  Grade 4 : White blood cell count decreased | 12
  Grade 3 : Neutrophil count decreased | 25
  Grade 4 : Neutrophil count decreased | 34
  Grade 3 : Lymphocyte count decreased | 6
  Grade 4 : Lymphocyte count decreased | 63
  Grade 3 : Haemoglobin decreased | 5
  Grade 3 : Platelet count decreased | 3
  Grade 4 : Platelet count decreased | 2

ADVERSE EVENTS:
Groups:
- SyB L-0501＋Rituximab: Drug: SyB L-0501
  A dose of 90 mg/m^2/day of SyB L-0501 is administered on Day 1 and Day 2 as an IV drip infusion, followed by 26-day observation. This is 1 cycle (28 days), which will be repeated for a maximum of 6 times.
  Drug: rituximab
  A dose of 375 mg/m^2 of rituximab is administered on Day 1 (Day 0 in Cycle 1 only) as an IV drip infusion, followed by 26-day observation. This is 1 cycle (28 days), which will be repeated for a maximum of 6 times. From Cycle 2, rituximab will be coadministered with SyB L-0501 on Day 1. However, if the investigator or sub-investigator judges that the coadministration is difficult, rituximab may be administered on Day 0.
Arm/Group | SyB L-0501＋Rituximab
Serious Adverse Events (participants affected / at risk) | 9/69
Other Adverse Events (participants affected / at risk) | 69/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SyB L-0501＋Rituximab (N=69)
Febrile neutropenia (Blood and lymphatic system disorders) | 3
tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
pneumonia cytomegaloviral (Infections and infestations) | 1
dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
cytogenetic abnormality (Congenital, familial and genetic disorders) | 1
atrial tachycardia (Cardiac disorders) | 1
pyrexia (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SyB L-0501＋Rituximab (N=69)
Anaemia (Blood and lymphatic system disorders) | 24
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 3
Lymphadenitis (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 3
Ventricular arrhythmia (Cardiac disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
External ear inflammation (Ear and labyrinth disorders) | 1
Steroid withdrawal syndrome (Endocrine disorders) | 1
Asthenopia (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 2
Dry eye (Eye disorders) | 1
Erythema of eyelid (Eye disorders) | 1
Scintillating scotoma (Eye disorders) | 1
Trichiasis (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Anal fissure (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 4
Colitis ischaemic (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 45
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 11
Dyspepsia (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 46
Oesophageal pain (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 13
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 6
Chills (General disorders) | 1
Fatigue (General disorders) | 6
Injection site bruising (General disorders) | 1
Injection site induration (General disorders) | 1
Injection site pain (General disorders) | 8
Injection site phlebitis (General disorders) | 1
Injection site reaction (General disorders) | 8
Local swelling (General disorders) | 1
Malaise (General disorders) | 37
Oedema (General disorders) | 3
Oedema peripheral (General disorders) | 3
Pain (General disorders) | 2
Pyrexia (General disorders) | 17
Thirst (General disorders) | 1
Injection site swelling (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Infusion site extravasation (General disorders) | 1
Injection site vasculitis (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 5
Liver disorder (Hepatobiliary disorders) | 1
Gallbladder polyp (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 2
Drug hypersensitivity (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 3
Hypogammaglobulinaemia (Immune system disorders) | 1
Sarcoidosis (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Chronic sinusitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 2
Cytomegalovirus infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Hepatitis viral (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 14
Oral candidiasis (Infections and infestations) | 2
Paronychia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 2
Cytomegalovirus viraemia (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Acarodermatitis (Infections and infestations) | 1
Aspergillus infection (Infections and infestations) | 1
Arthropod sting (Injury, poisoning and procedural complications) | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 28
Thermal burn (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 18
Amylase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 22
Beta 2 microglobulin increased (Investigations) | 3
Blood albumin decreased (Investigations) | 5
Blood bilirubin increased (Investigations) | 3
Blood creatinine increased (Investigations) | 5
Blood immunoglobulin A decreased (Investigations) | 21
Blood immunoglobulin G decreased (Investigations) | 21
Blood immunoglobulin M decreased (Investigations) | 32
Blood lactate dehydrogenase increased (Investigations) | 22
Blood potassium decreased (Investigations) | 1
Blood urea increased (Investigations) | 1
Blood uric acid increased (Investigations) | 3
C-reactive protein increased (Investigations) | 18
CD4 lymphocytes decreased (Investigations) | 64
Electrocardiogram QT prolonged (Investigations) | 2
Eosinophil count increased (Investigations) | 11
Gamma-glutamyltransferase increased (Investigations) | 15
Blood urine present (Investigations) | 1
Haemoglobin decreased (Investigations) | 7
Low density lipoprotein increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 67
Lymphocyte count increased (Investigations) | 1
Monocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 65
Neutrophil count increased (Investigations) | 9
Platelet count decreased (Investigations) | 38
Protein total decreased (Investigations) | 8
Protein urine (Investigations) | 1
Red blood cell count decreased (Investigations) | 9
Weight decreased (Investigations) | 9
Weight increased (Investigations) | 5
White blood cell count decreased (Investigations) | 69
White blood cell count increased (Investigations) | 6
Blood bilirubin decreased (Investigations) | 1
Neutrophil percentage decreased (Investigations) | 1
Neutrophil percentage increased (Investigations) | 1
Electrocardiogram ST-T segment abnormal (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 13
Occult blood (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 4
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 30
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 3
Dizziness postural (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 13
Headache (Nervous system disorders) | 12
Neuropathy peripheral (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Sensory disturbance (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Lacunar infarction (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 19
Haematuria (Renal and urinary disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 3
Urinary retention (Renal and urinary disorders) | 1
Breast swelling (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 6
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Acne (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Miliaria (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 13
Rash (Skin and subcutaneous tissue disorders) | 29
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Urticaria (Skin and subcutaneous tissue disorders) | 2
Xeroderma (Skin and subcutaneous tissue disorders) | 1
Tooth extraction (Surgical and medical procedures) | 1
Flushing (Vascular disorders) | 4
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Orthostatic hypotension (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 4
Vascular pain (Vascular disorders) | 11
Vasculitis (Vascular disorders) | 20
Hot flush (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No